CLINICAL TRIAL: NCT04753333
Title: Efficacy of Electromyographic-biofeedback Supplementation Training on Quadriceps Strengthening With Patellar Taping in Patellofemoral Pain Syndrome Among Young Adult Male Athletes
Brief Title: Quadriceps Strengthening With Patellar Taping in Patellofemoral Pain Syndrome Among Young Adult Male Athletes
Acronym: PFPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, Shahnaz Hasan, PhD, Associate Professor, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSRMajmaahU; 2020-26 (Other Grant/Funding Number: DSR)
Record Dates: First submitted 2021-01-22; First posted 2021-02-15 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Patellofemoral Disorder; Anterior Knee Pain
Keywords: Pain; Strength; Function; PFPS; Athletes; Young adults
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Experimental: Participants in this group will receive electromyography biofeedback (EMG-BF) guided strength training along with patellar taping
  No Intervention: Control: Participants in this group will receive Sham EMG-BF guided strength training without patellar taping
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The participants in the experimental group will receive Electromyographic-biofeedback guided (EMG-BF) isometric quadriceps strengthening with patellar taping five days a week for four weeks.
  Interventions: Behavioral: Electromyography biofeedback (EMG-BF)
- Control (Placebo Comparator): The participants in the experimental group will receive Sham EMG-BF guided isometric quadriceps strengthening without patellar taping five days a week for four weeks.
  Interventions: Behavioral: Sham electromyography biofeedback (EMG-BF)

INTERVENTIONS:
Behavioral: Electromyography biofeedback (EMG-BF) — Participants in this group will receive electromyography biofeedback (EMG-BF) guided strength training with patellar taping
  Other Names: Patellar Taping
  Arms: Experimental
Behavioral: Sham electromyography biofeedback (EMG-BF) — Participants in this group will receive Sham electromyography biofeedback (EMG-BF) guided strength training without patellar taping
  Arms: Control

SUMMARY:
This study aims to investigate the effects of electromyography biofeedback (EMG-BF) guided isometric quadriceps strengthening with patellar taping and isometric exercise alone in young adult male athletes with patellofemoral pain syndrome (PFPS).

DETAILED DESCRIPTION:
A total of 60 adult male athletes aged 18 to 45 years will be recruited from two cities (Majmaah and Riyadh) of Saudi Arabia. Subjects will be included with the history of knee pain during activities such as descending and ascending stairs, squatting, and running, had positive J sign (lateral tilt of patella), and a sign of patellar malalignment on the radiograph. Individuals with the history of fracture around knee, patella dislocation, knee deformity (e.g., genu varum), flexion contracture, ligaments/meniscal injuries, and osteoarthritis of knee will be excluded from the study. The protocol was submitted to and approved by the ethical sub-committee of College of applied medical science, Majmaah, Saudi Arabia (Ethics number: MUREC-Nov./COM-2O20/11-2). Participants will be requested to sign a written informed consent form approved by the institution ethics committee.

Participants will be randomly assigned to Group A (experimental group): electromyography biofeedback (EMG-BF) guided maximum voluntary isometric contraction exercise with patellar taping; Group B (control group): sham EMG-BF guided maximum voluntary isometric contraction without patellar taping. The outcome measure for this study will be the mean changes in maximum voluntary isometric contraction (MVIC) of the quadriceps muscle, pain intensity, and functional status up to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Knee pain during activities such as descending and ascending stairs, squatting, and running,
2. Positive J sign (lateral tilt of patella),
3. Sign of patellar malalignment on radiograph.

Exclusion Criteria:

1. Fracture around knee,
2. Patella dislocation,
3. Knee deformity (e.g., genu varum),
4. Knee flexion contracture,
5. Ligaments/meniscal injuries, and
6. Osteoarthritis of knee.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Mean changes in pain intensity | up to 6 weeks
  The 10-cm visual analogue scale (VAS) will be used for the assessment of pain intensity. Each participant will be instructed to report their current intensity of pain on a 10-cm scale between two anchors 0 (indicates no pain) and 10 (indicates maximum pain).
Mean changes in knee function | up to 6 weeks
  Knee function will be assessed using the validated Anterior Knee Pain scale. It comprised of 13 questions designed to evaluate difficulties related to PFPS such as presence of a limp, walking ability, need for support, squatting, stair climbing, jumping, running, pain, abnormal painful kneecap movement, prolonged sitting with knees flexed, atrophy of the thigh, swelling, and flexion deficiency. Total scores range between 0 and 100. A higher score suggests lower symptoms and better functional capacity.
Mean changes in quadriceps muscle strength | up to 6 weeks
  Maximum voluntary isometric strength of quadriceps femoris muscle will be measured using an isokinetic dynamometer. Participants will be made in a sitting position and secured using the stabilization straps with the knee joint in 60 degrees of flexion, as this position has resulted in the most significant torque output. They will be verbally encouraged to carry out three maximal voluntary isometric contractions of quadriceps with 5-sec rest. The best of the three maximum peak torque will be used for the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Shahnaz Hasan, PhD, Principal Investigator — Majmaah University
Locations (1):
- Physiotherapy & Rehabilitation center, Al Majma'ah, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Data will be kept secure with the principal investigator (Dr. Asma Alonazi) and sub-investigator (Dr. Shahnaz Hasan) due to confidentiality issues